CLINICAL TRIAL: NCT06352567
Title: A View of Perceived Symptoms Associated with Chemotherapy-Induced Peripheral Neuropathy in Patients with Breast Cancer
Brief Title: Symptoms Associated with Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Alper Tuğral, Principal Investigator, Izmir Bakircay University
Other Study IDs: BakircayU1394/1414
Record Dates: First submitted 2024-03-29; First posted 2024-04-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Breast Cancer; Breast Cancer Female
Keywords: Breast Cancer; Neuropathy; Chemotherapeutic Toxicity; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast Cancer: Patients diagnosed with breast cancer who underwent systemic adjuvant or neoadjuvant chemotherapy will be assessed with the European Organization for Research and Treatment of Cancer-Chemotherapy Induced Peripheral Neuropathy (EORTC-CIPN20) questionnaire within completion of the systemic chemotherapy in 1-2 months.
  Interventions: Other: European Organization for Research and Treatment of Cancer-Chemotherapy Induced Peripheral Neuropathy (EORTC-CIPN20) questionnaire

INTERVENTIONS:
Other: European Organization for Research and Treatment of Cancer-Chemotherapy Induced Peripheral Neuropathy (EORTC-CIPN20) questionnaire — It consists of a total of 20 items each is scored from "1: not at all" to "4: very much" in a 4-point Likert scale. Individuals are requested to fill out by considering their last week. Sensory, motor, and autonomic subscales are reported within its constructs. A total of 9, 8, and 3 items are referred to as sensory, motor, and autonomic disturbances, respectively

SUMMARY:
Breast cancer remains the most frequent type of cancer globally. Nevertheless, the increased rate of disease-free survival of breast cancer brought the specific need of managing of short and long-term side effects of multimodal treatment. Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most debilitating conditions which is characterized by a wide variety of experienceable symptoms by patients that need to be addressed in detail. Therefore, in this cross-sectional study, it was aimed to assess the potential symptoms associated with CIPN of patients with breast cancer who underwent systemic chemotherapy. In addition, it was aimed to assess the potential associations between experienced symptoms of CIPN and sociodemographic (age, body mass index etc.) and clinical features (mean exposed dose, type of surgery (if any) etc.).

DETAILED DESCRIPTION:
Patients with breast cancer who underwent systemic chemotherapy were assessed with the European Organization for Research and Treatment of Cancer-Chemotherapy Induced Peripheral Neuropathy (EORTC-CIPN20) questionnaire within 1-2 months after completion of systemic chemotherapy. A simple data form was implemented in which patients' age, weight, height, marital status, smoking status, etc were investigated. In addition, the dose of the exposure of systemic chemotherapy was calculated according to the Body Surface Area (BSA) and DuBois formulation as follows: BSA [m2] = Weight [kg]0.425 × height (cm)0.725 × 0.007184]. The universal dose calculations were used to calculate the mean exposure according to the following doses for each patient-specific to their chemotherapy regimen: Four cycles of Anthracycline were applied 14 days apart 60 mg/m2 intravenous (IV), 12 cycles of Paclitaxel were applied seven days apart 80 mg/m2 IV, and four cycles of Docetaxel were applied 21 days apart 75 mg/m2 IV.

ELIGIBILITY:
Inclusion Criteria:

* Being a volunteer to participate
* aged over 18 years old
* being female
* being a candidate for systemic chemotherapy

Exclusion Criteria:

* Having distant metastasis
* Having comorbidities that might contribute to or cause sensorial and motor deficits such as multiple sclerosis, diabetes, polyneuropathy, etc.,
* Prolonged surgical (if any) complications (i.e. pain, seroma, etc.)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being female.
Study Population: Patients who were diagnosed with breast cancer and referred to the medical oncology unit for the purpose of systemic chemotherapy treatment were screened and invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Assessment of perceived Chemotherapy Induced Peripheral Neuropathy symptoms | From completion of systemic chemotherapy up to two months
  European Organization for Research and Treatment of Cancer-Chemotherapy Induced Peripheral Neuropathy (EORTC-CIPN20) questionnaire was used to assess symtomps associated with CIPN. Higher scores indicate worse, or vice versa. Minimum and maximum score are 0 and 100, respectively. The questionnaire is calculated in three different sub-domains as follows: Autonomic, sensory and motor.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Tuğral, Ph.D., Principal Investigator — Izmir Bakircay University; Murat Akyol, MD, Prof., Study Director — Izmir Bakircay University
Locations (1):
- Bakircay University Çiğli State and Training Hospital, Department of Medical Oncology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tugral A, Aribas Z, Akyol M, Bakar Y. Assessment of sensorimotor and strength related function of breast cancer patients during systemic drug therapy: a prospective observational study. BMC Cancer. 2023 Oct 14;23(1):981. doi: 10.1186/s12885-023-11494-x. PMID 37838686
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Zhi WI, Chen P, Kwon A, Chen C, Harte SE, Piulson L, Li S, Patil S, Mao JJ, Bao T. Chemotherapy-induced peripheral neuropathy (CIPN) in breast cancer survivors: a comparison of patient-reported outcomes and quantitative sensory testing. Breast Cancer Res Treat. 2019 Dec;178(3):587-595. doi: 10.1007/s10549-019-05416-4. Epub 2019 Aug 27. PMID 31456070
- [Background] Molinares D, Kurtevski S, Zhu Y. Chemotherapy-Induced Peripheral Neuropathy: Diagnosis, Agents, General Clinical Presentation, and Treatments. Curr Oncol Rep. 2023 Nov;25(11):1227-1235. doi: 10.1007/s11912-023-01449-7. Epub 2023 Sep 13. PMID 37702983
- [Background] Song SJ, Min J, Suh SY, Jung SH, Hahn HJ, Im SA, Lee JY. Incidence of taxane-induced peripheral neuropathy receiving treatment and prescription patterns in patients with breast cancer. Support Care Cancer. 2017 Jul;25(7):2241-2248. doi: 10.1007/s00520-017-3631-x. Epub 2017 Feb 16. PMID 28204996